CLINICAL TRIAL: NCT05603897
Title: Utility of Non-standardized Clinical Swallow Evaluation vs. Standardized Swallow Evaluation to Identify the Presence of Dysphagia and Risk for Aspiration in Patients Post-ischemic Stroke in Acute Inpatient Rehabilitation
Brief Title: Non-standardized vs. Standardized Screening for Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gemayaret Alvarez, Attending Physician, University of Miami
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20220558
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dysphagia
Keywords: difficulty swallowing
MeSH Terms: conditions — Deglutition Disorders | interventions — methyl N-acetylsibirosaminide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mann Assessment of Swallowing Ability (MASA) Group (Experimental): Participants in this group will receive the MASA dysphagia screening once upon admission to inpatient rehabilitation for approximately 20 minutes.
  Interventions: Other: Mann Assessment of Swallowing Ability (MASA) (dysphagia screening tool)
- Non-standardized clinical swallow evaluation Group (Other): Participants in this group will receive standard of care treatment (dysphagia screening once upon admission to inpatient rehabilitation using a non-standardized clinical swallow evaluation for approximately 15 minutes).
  Interventions: Other: Non-standardized clinical swallow evaluation

INTERVENTIONS:
Other: Mann Assessment of Swallowing Ability (MASA) (dysphagia screening tool) — Upon 1-2 days of admission to inpatient rehabilitation, the MASA will be administered for approximately 20 minutes during initial speech language pathology evaluation. The MASA will be administered at bedside as a cognitive/speech language evaluation as well as oropharyngeal function examination.
  Arms: Mann Assessment of Swallowing Ability (MASA) Group
Other: Non-standardized clinical swallow evaluation — Participants will receive current standard of care for dysphagia screening and treatment.
  Arms: Non-standardized clinical swallow evaluation Group

SUMMARY:
The purpose of this study is to compare two different screening tests for detecting dysphagia (difficulty swallowing) as well as the risk for aspiration (silent swallowing of liquids/solids into the lungs) in patients after an ischemic stroke (when a blood clot blocks or narrows an artery leading to the brain).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Patients admitted to Lynn Rehabilitation Center with an admitting diagnosis consistent with acute ischemic stroke within the past 1 month
* Patients able to provide informed, written consent. If patients are not cognitively able to give informed consent, then consent will be obtained from patient proxy in person or over the phone
* Able to read and comprehend verbal instruction in English and/or Spanish

Exclusion Criteria:

* Adults > 80 years old
* Pregnant women
* Prisoners
* Those with a prior history of dysphagia
* Those with any diagnoses that include acute intracranial hemorrhage, subdural hematoma, subarachnoid hemorrhage, traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Dysphagia measured by MASA | Up to 20 minutes
  The MASA is a 24-item clinical test that evaluates swallowing in the order in which swallowing phases occur. Each item is quantitatively scored using either a 5-point or 10-point score at the end of which a total score out of 200 is summed up. The MASA takes approximately 15-20 minutes to perform and can then be repeated during a patient's clinical course to monitor for recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Gemayaret Alvarez, MD, Principal Investigator — University of Miami
Locations (1):
- Lynn Rehabilitation Center / University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No